CLINICAL TRIAL: NCT00004789
Title: Phase I/II Study of Heme Arginate and Tin Mesoporphyrin for Acute Porphyria
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11887; UTMB-398
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Porphyria
Keywords: inborn errors of metabolism; acute porphyria; rare disease
MeSH Terms: conditions — Porphyrias; Metabolism, Inborn Errors; Porphyria, Acute Intermittent; Rare Diseases | interventions — heme arginate; tin mesoporphyrin

INTERVENTIONS:
Drug: heme arginate
Drug: tin mesoporphyrin

SUMMARY:
OBJECTIVES: I. Evaluate the efficacy and safety of heme arginate in the treatment of 20 patients with acute attacks of porphyria.

II. Evaluate the efficacy and safety of heme arginate in preventing frequent exacerbations of acute porphyria in up to 15 patients.

III. Estimate the lowest effective dose of heme arginate (0.3, 1.0, or 3.0 mg/kg) in reducing porphyrin precursors in 12 stable patients with acute intermittent porphyria in remission.

IV. Evaluate the safety and efficacy of tin mesoporphyrin used in combination with heme arginate in reducing porphyrin precursors in 12 stable patients with acute intermittent porphyria in remission.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This project involves 4 studies: an unblinded multicenter treatment study, an unblinded prevention study, a controlled dose-ranging study, and a controlled drug combination dose-ranging study.

In the treatment study, participants with acute attacks of porphyria receive intravenous heme arginate daily for 4 days. Treatment may be extended to 7 days in patients with severe attacks and slow recovery; these data are analyzed separately.

In the prevention study, participants receive weekly infusions of heme arginate for 6 months. Treatment may be extended in selected cases; these data are analyzed separately. If an acute attack occurs, patients are treated with a standard course of heme arginate. Participants are followed weekly for 6 months after preventive treatment.

In the dose-ranging study, 4 groups of 3 patients are randomly assigned to standard and low-dose heme arginate infusions, administered daily for 4 days. After a washout of 4-12 weeks, patients are crossed to a second dose. In 2 of the 4 groups, patients cross between heme arginate and a normal saline control.

In the combination dose-ranging study, 4 groups of 3 patients are randomly assigned to 1 of 2 doses of tin mesoporphyrin. After a 4-12 week washout, these patients are crossed to a standard or low-dose heme arginate infusion. After a second 4-12 week washout, patients are given a combination infusion of tin mesoporphyrin followed by heme arginate.

All participants are given a special diet to prevent fluctuations in porphyrin precursors.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Well-documented acute porphyria, i.e.: Acute intermittent porphyria Variegate porphyria Hereditary coproporphyria

--Patient Characteristics--

* No pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59
Dates: Start 1993-07

CONTACTS AND LOCATIONS:
Overall Officials: Karl Elmo Anderson, Study Chair — University of Texas